CLINICAL TRIAL: NCT05297747
Title: Is Adrenomedullin Upregulation Due to Apical Periodontitis Independent of Periodontal Disease?
Brief Title: Adrenomedullin Upregulation in Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Principal Investigator, Clinical Associate Professor, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 472-10.06.2020
Record Dates: First submitted 2022-03-09; First posted 2022-03-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Periapical Periodontitis
Keywords: Apical periodontitis, Chronic periodontitis, Mid regional proadrenomedullin, IL-12, TNF-α
MeSH Terms: conditions — Periapical Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apical periodontitis (Experimental): Radiography of the patients in the apical periodontitis group was evaluated and blood samples were collected from those patients
  Interventions: Diagnostic Test: Apical periodontitis
- Chronic periodontitis (Experimental): Radiography of the patients in the chronic periodontitis group was evaluated and blood samples were collected from those patients
  Interventions: Diagnostic Test: Chronic periodontitis
- Control (No Intervention): Radiography of the participants in the healthy, control group was evaluated and blood samples were collected from those participants

INTERVENTIONS:
Diagnostic Test: Apical periodontitis — Radiography of the patients were taken. Blood samples were collected from those patients.
  Arms: Apical periodontitis
Diagnostic Test: Chronic periodontitis — Radiography of the patients were taken. Blood samples were collected from those patient
  Arms: Chronic periodontitis

SUMMARY:
The aim of the present study was to investigate the relationship between Apical periodontitis (AP) severity and inflammatory markers (IL-12, TNF-alpha), and Mid-Regional Pro Adrenomedullin (MR-proADM) in patients with AP. A total of 174 subjects were divided into three categories: AP group (n=82), Chronic periodontitis (CP) group (n=42), healthy control group (n=50). Blood samples were collected from all of the patients. Enzyme-linked immunosorbent assay was used to evaluate the samples.

DETAILED DESCRIPTION:
Bone destruction in apical periodontitis (AP) depends on the microorganisms' efficiency to breach the host-epithelial barrier and various antimicrobial peptides. Mid-regional pro adrenomedullin (MR-proADM) is one such potent antimicrobial peptide, which plays a regulatory and stabilizing role among proinflammatory and anti-inflammatory cytokines. A broad range of cells and tissues produce MR-proADM such as adrenal medulla, kidney, lungs, and endothelial cells. MR-proADM was found to be present in circulation and in various biological fluids. It is reported to function both as a generalized hormone and locally affecting autocrine or paracrine mediator. Its plasma level is usually elevated in certain conditions such as heart failure, hypertensive situations, cerebro-vascular events, chronic kidney failure, diabetes mellitus, sepsis and periodontitis. Besides these, MR-proADM has drawn attention as it stimulates the proinflammatory cytokine IL-6 and suppresses cytokines, like TNF- α, for regulating inflammation, being a potent of inhibitor of apoptosis and stimulating angiogenesis in tumor cells. However, there is still a large information gap on MR-proADM. Despite all these effects, there is not enough information in the literature about the effect of MR-proADM on oral and dental health and its effectiveness in apical periodontitis. Whether AP can cause any alterations in the MR-proADM value is also unknown.

Therefore, the aim of this study is to investigate the relationship between AP severity and inflammatory markers (IL-12, TNF-alpha), and MR-proADM in patients with AP. In addition, the results will be compared with the results of healthy controls and patients with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

Must be systemically healthy Patients with only apical periodontitis (for AP group) Patients with only chronic periodontitis (for CP group) Orally healthy patients

Exclusion Criteria:

any local or systemic inflammatory disease connective tissue diseases like systemic lupus erythematosus (SLE) cardiovascular disease inflammatory and rheumatic disease diabetes rheumatoid arthritis, or Behcet's disease granulomatous diseases like sarcoidosis inflammatory intestinal diseases like ulcerative colitis and Crohn's autoimmune intestinal diseases like celiac thyroid diseases like Hashimoto and Graves patients who had taken antibiotics and/or anti-inflammatory drugs within the last 6 months those with pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Mid-Regional Pro Adrenomedullin levels | through study completion, an average of 1 year
  Biomarker levels of all patients were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After publication of the study, we are planning to share our data
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: by email